CLINICAL TRIAL: NCT00175994
Title: Bioavailability and Metabolism of Voriconazole as a Function of the CYP2C19 Genotype
Brief Title: Bioavailability and Metabolism of Voriconazole in Relation to Its Modulation by the CYP2C19 Genetic Polymorphism
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Other Study IDs: 2005-001649-41; K117
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-04-17 (Estimated); Status verified 2007-04

CONDITIONS: Healthy
Keywords: voriconazole; genotype; bioavailability; metabolic clearance

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purposes of this study are:

* To determine the absolute bioavailability of voriconazole after a single oral dose (400 mg voriconazole [VFEND brand]) in comparison to intravenous (i.v.) administration (400 mg VFEND, equivalent to two 10 mg/ml-infusates, each containing 200 mg voriconazole [VRC]) in healthy individuals stratified according to the three predominant CYP2C19 genotypes
* To investigate the possible pathways of metabolism and their modulation according to genetic polymorphism of CYP2C19 after i.v. and oral administration of VRC.

DETAILED DESCRIPTION:
As CYPs are mainly involved in VRC metabolism it is likely that also gut wall metabolism by CYPs occurs. However, no substantial first pass metabolism of VRC has been reported. In humans the VRC metabolism has not been studied systematically. It is therefore important to assess VRC metabolism on its own and in addition the influence of CYP2C19 genetic polymorphisms on the formation of the different VRC metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Good state of health (physically and mentally)

Exclusion Criteria:

* Any regular drug treatment within the last two months except for oral contraceptives in female participants
* Any intake of a substance known to induce or inhibit drug metabolising enzymes or transport system enzymes within a period of less than 10 times the respective elimination half-life
* Any acute or chronic illness or clinically relevant findings in the pre-study examination
* Allergies (except for mild forms of hay fever) or history of hypersensitivity reactions
* Smoking (regular or irregular)
* Excessive alcohol drinking (more than approximately 30 g alcohol per day)
* Positive drug screening or known or admitted drug abuse

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2005-07; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Mikus, MD BSc, Principal Investigator — Department Internal Medicine VI
Locations (1):
- Clinical Research Unit, Department Internal Medicine VI, Heidelberg, Germany